CLINICAL TRIAL: NCT02810600
Title: Phase II Study to Measure the Safety of 68Ga-DOTA-TATE PET/CT in the Diagnosis of Tumors Expressing Somatostatin Receptors
Brief Title: Study to Measure the Safety of 68Ga-DOTA-TATE PET/CT in the Diagnosis of Tumors Expressing Somatostatin Receptors
Acronym: PET/Ga68
Status: Completed | Type: Observational
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: Gallium DOTATATE/PET scan
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Gallium-68 DOTA TATE PET scan — One PET/CT scan using Gallium-68 DOTA TATE

SUMMARY:
Phase-II, prospective, open label, no control group to assess the safety of 68Ga-DOTA-TATE injection in patients with suspected or diagnosed with tumors expressing somatostatin receptors. Each included patient will receive an administered dose of 50 mcg or less of the peptide (DOTA-TATE) and a range of activity between 100 - 200 MBq of 68Ga-DOTA-TATE.

The efficacy of 68Ga-DOTA-TATE in assessing this kind of tumors has been proved by numerous studies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected or proven tumors expressing Somatostatin receptors
2. Informed consent by patient (or parents if patient is less than 18 years of age)

Exclusion Criteria:

1. Pregnancy (confirmed). In the case of a diagnostic procedure in a patient who is or may be pregnant, a clinical decision is necessary considering the benefits against the possible harm of carrying out any procedure.
2. Patient refusal to participate.
3. Impossibility to tolerate a decubitus position for 25 minutes
4. Prior allergic reaction to DOTA-TATE or somatostatin analogs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected or diagnosed with tumors expressing somatostatin receptors
Sampling Method: Non-Probability Sample
Enrollment: 2120 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Record all adverse events | June 2016-June 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No